CLINICAL TRIAL: NCT06051591
Title: Food FARMacia: Reducing Childhood Obesity in Households With Food Insecurity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jennifer Woo Baidal, Associate Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 76726; R01DK134463 (NIH)
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Nutrition, Healthy
Keywords: Childhood Obesity; Food Insecurity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized and assigned to enroll in the Food FARMacia program for the duration of the study period or to receive usual care.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will not be masked as they will be receiving twice monthly groceries if they are enrolled in the Food FARMacia program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control (Active Comparator): Participants will receive nutrition education and anticipatory guidance to support healthy meal preparation in addition to usual care.
  Interventions: Behavioral: Self-directed meal preparation support
- Food FARMacia intervention (Experimental): Participants will enroll in the Food FARMacia program and receive groceries twice monthly for 6 months. They will also receive nutrition education and anticipatory guidance to support healthy meal preparation.
  Interventions: Behavioral: Food FARMacia Program; Behavioral: Self-directed meal preparation support

INTERVENTIONS:
Behavioral: Food FARMacia Program — Twice monthly delivery of groceries with about 12 meals per household member for up to 4 household members for 6 months.
  Arms: Food FARMacia intervention
Behavioral: Self-directed meal preparation support — Nutrition education and anticipatory guidance to support healthy meal preparation

SUMMARY:
The goal of this clinical trial is to test whether the Food FARMacia intervention to reduce food insecurity is feasible and accepted among families with an infant age 6 to less than 18 months receiving pediatric primary care.

All participants will receive nutrition education and anticipatory guidance to support healthy meal preparation in addition to usual care.

DETAILED DESCRIPTION:
Childhood obesity remains highly prevalent and originates early in life. Efficacious early life interventions to prevent childhood obesity are lacking, particularly among populations most burdened by childhood obesity. Food insecurity - defined as lack of enough food for an active, healthy life - may play key upstream roles in etiologies of obesity through establishment of unhealthy dietary patterns and stress-related metabolic perturbations. Household food insecurity during the first 24 months of life is a risk factor for later childhood obesity. Professional organizations recommend integration of household food insecurity screening into routine pediatric primary care. Yet, a critical gap exists in identification of efficacious clinical interventions to reduce food insecurity. Another gap exists in understanding relationships between food insecurity and etiologies of obesity. Food FARMacia is a clinically based mobile food pantry intervention developed to address the high prevalence of food insecurity among pediatric patients. No randomized trials of a clinically-based mobile food pantry intervention in pediatric primary care exist. To understand the role of food insecurity in etiologies of childhood obesity, efficacious interventions to reduce food insecurity are needed.

Household food insecurity during infancy is a risk factor for later childhood obesity. In this pilot and feasibility study, the investigators will randomly assign infants and their parent in households with food insecurity to either 1) the Food FARMacia mobile food pantry intervention with twice monthly food distributions and self-directed meal preparation support or 2) self-directed meal preparation support. Infants age 6 to <18 months who are patients at Stanford University/Stanford Health Care who screen positive for food insecurity will potentially be eligible participants for recruitment. Parents will be asked to respond to survey questions about health behaviors for themself and their infant at baseline and follow-up.

The investigators will measure vital signs (e.g., weight and height/length) for parents and infants at baseline and follow-up. The investigators will examine feasibility, acceptability, and satisfaction with the study procedures and intervention materials. The investigators will estimate intervention effects on infant weight characteristics and explore potential mediators such as reduction in food insecurity and changes in nutrition and other established obesity risk factors to inform a subsequent full-scale trial. If successful, results will lead to a full-scale trial to test effects of the intervention on food insecurity, nutrition, and infant growth. Eventually, these study results could transform clinical care to reduce childhood obesity.

ELIGIBILITY:
Inclusion Criteria for Child:

* Age 6 to < 18 months at enrollment
* Born gestational age 37 weeks or later without evidence of undernutrition at routine health care visits
* In household with food insecurity at time of screening phone call based on an affirmative response on the 2-item Hunger Vital Signs™ screening tool
* Primary pediatric care patient at Stanford University/Stanford Health Care Network
* Planned continuation of primary pediatric care at Stanford University/Stanford Health Care
* Living in a community setting (not inpatient or living in a nursing/long-term care setting) with a caretaker enrolled in this study

Exclusion Criteria for Child:

* Gestational age < 37 weeks
* Small-for-gestational age at birth (birth weight for gestational age less than 10th percentile)
* Weight-for-length < 3rd percentile
* Body Mass Index < 5th percentile for age and sex
* Children in household previously enrolled in this study or the Food FARMacia program
* Conditions that substantially interfere with growth or mobility (e.g., complex congenital heart disease, cystic fibrosis)
* Children with special diets (e.g., tyrosinemia, enteral tube feeding)
* Children with chronic diseases that interfere with nutrition and growth as determined by investigators

Inclusion Criteria for Parent/Legal Guardian:

* Primary caretaker of infant eligible for study and with planned enrollment in this study
* Age 18 years or older
* Ability to respond to questions in English and/or Spanish
* Willing for self and infant to be randomized into a RCT and complete all study components
* Gives permission to receive messages to their mobile device, email, and or place of residence
* Gives permission to complete all study procedures for self and infant
* Capable of providing informed consent for self and infant

Exclusion Criteria for Parent/Legal Guardian:

* Pregnancy at baseline visit because of unique nutritional needs
* Age < 18 years at baseline because of unique developmental differences of adolescents and New York State regulations
* Inability to complete study visits or intervention components
* Unwillingness or inability to commit to a 6-month research study for self or infant
* Unable to give informed consent
* Underlying disease/treatment that might interfere with participation in/completion of the study (e.g., significant gastrointestinal conditions, major psychiatric disorders, and others at the discretion of the study clinician)

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility | 24 months
  Completion of enrollment of 80 households within the study timeframe
Retention Rate | 6 months
  At least 70% with complete follow-up visits at 6-month follow-up
Attendance Rate (Proportion of food distributions attended/received) - Intervention Arm | 6 months
  At least 70% median attendance rate for twice monthly food distributions at 6-month follow-up
Intervention Satisfaction - Intervention Arm | 6 months
  Average report of agree or strongly agree (mean score 4 or higher on a 5-point scale) with intervention satisfaction at 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Woo Baidal, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant level data
Supporting Information: Study Protocol
Time Frame: Beginning 3 months after peer-reviewed publication and up to 36 months after publication.
Access Criteria: Investigators who provide a proposal for data use that is approved by the study investigators. Information on submitting proposals and accessing data may be obtained by emailing the study PI and coordinator. A signed data use agreement will be required.